CLINICAL TRIAL: NCT00159003
Title: Molecular Analysis of Genetic Elements Which May Influence Predisposition and Prognosis of Hematological Malignancies in Different Ethnic Groups in Israel
Brief Title: Analysis of Genetic Factors Related to Predisposition and Prognosis of Hematological Malignancies in Israel
Status: Completed | Type: Observational
Sponsor: Deborah Rund (Other)
Responsible Party: Sponsor-Investigator, Deborah Rund, Senior Hematologist, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Other Study IDs: 132910-HMO-CTIL
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Acute Myeloid Leukemia; Chronic Lymphocytic Leukemia; Chronic Myelogenous Leukemia
Keywords: drug metabolism and disposition enzymes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA only
Oversight: Data Monitoring Committee: No

SUMMARY:
There are naturally occuring variations in the genetic makeup of all of us. Some of these variations may contribute to a change in susceptibility toward different diseases or change the prognosis.

We are studying these genetic variations in patients with leukemia. The genes we are studying are those which influence detoxification of drugs and toxins.

DETAILED DESCRIPTION:
We have prepared DNA on patients with leukemia (AML, CML and CLL) and we are studying the influence of polymorphisms in drug metabolism and disposition genes on predisposition and prognosis of these types of leukemia. The genes we are studying include: MDR1, CYP3A4, NQO1, NAT1/2, GST, hOCT. We plan to study other genes that may be contributory.

Study includes comparing the frequency of polymorphisms in these genes with the frequency in the general population and the study of DNA biding proteins which bind at the sites of these polymorphisms.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of acute myeloid leukemia or chronic lymphocytic leukemia

Exclusion Criteria:

* under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Hadassah Hospital with AML or CLL.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 1998-01-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah G Rund, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Chanock S. Genetic variation and hematology: single-nucleotide polymorphisms, haplotypes, and complex disease. Semin Hematol. 2003 Oct;40(4):321-8. doi: 10.1016/s0037-1963(03)00198-7. PMID 14582082